CLINICAL TRIAL: NCT07230483
Title: An Open-Label, Multicenter Study to Evaluate Long-Term Safety and Efficacy of CM512 in Atopic Dermatitis Patients.
Brief Title: A Long-term Safety and Efficacy Study Evaluating CM512 in Atopic Dermatitis.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM512-101103
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental)
  Interventions: Biological: CM512
- Group 2 (Experimental)
  Interventions: Biological: CM512
- Group 3 (Experimental)
  Interventions: Biological: CM512
- Group 4 (Experimental)
  Interventions: Biological: CM512

INTERVENTIONS:
Biological: CM512 — CM512 subcutaneous injection

SUMMARY:
This is an Open-label ,Multicenter Study to evaluate Long-Term Safety and Efficacy of CM512 in patients with Atopic Dermatitis who have completed treatment in parent CM512 Study.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study and voluntarily sign a written informed consent form (ICF).
* Subjects who have completed the week 18 evaluation in the parent study CM512-101102 or the End of Study(EOS) visit in the parent study CM512-100001.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Any other condition assessed by the investigator that makes participants unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 52 weeks
  The incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China